CLINICAL TRIAL: NCT06439628
Title: A Chinese Real-world Study of Rimegepant for the Acute Treatment of Migraine
Brief Title: ARISE-A Chinese Real-world Study of Rimegepant for the Acute Treatment of Migraine
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Shengyuan Yu, Director, Chinese PLA General Hospital
Other Study IDs: 89127781
Record Dates: First submitted 2023-12-13; First posted 2024-06-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Rimegepant treatment group
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — patients take rimegepant to treat migraine attack as needed

SUMMARY:
Research question and objectives Primary endpoint

• To evaluate the effectiveness of Rimegepant in the acute treatment of migraine as measured by most severe pain, onset of pain relief, satisfaction with pain relief, and satisfaction with return to normal function post-dose.

Secondary Objectives

* To evaluate the effectiveness of Rimegepant in the acute treatment of migraine as measured by onset of associated symptoms relief.
* To evaluate the long-term effect of Rimegepant treatment on the treatment satisfaction and global impression of change at months 3，6 and 12.

Exploratory Objective

* To evaluate the long-term effectiveness of Rimegepant by evaluating the changes from baseline in any decrease in MMD with any intensity in those participants with baseline MMD ≥6 days.
* To evaluate the long-term effectiveness of Rimegepant by evaluating the changes from baseline of any decrease of MHD.
* To evaluate the long-term effectiveness of Rimegepant by evaluating any decrease of mean number of moderate to severe migraine days per month in those participants with baseline MMD ≥6 days
* To evaluate the changes from baseline in the percentage of MOH and chronic migraine transformation to episodic migraine during Rimegepant long-term (PRN) use.
* To evaluate the changes from baseline of Rimegepant usage, other migraine-related medication usage and MO during Rimegepant long-term (PRN) use.
* To evaluate the changes from baseline on quality of life, function, depression and anxiety at months 3, 6 and 12.
* To evaluate the association between the timing of Rimegepant dosing (dosing at pain free while with any prodrome symptoms/ dosing at pain free while with any aura symptoms / dosing at mild pain/ dosing at moderate pain/ dosing at severe pain) and the acute treatment effectiveness of Rimegepant.
* To evaluate the acute treatment effectiveness of Rimegepant in migraine participants with a history of insufficient response or intolerable to NSAIDs /Triptans /Combination analgesic.
* To evaluate the acute treatment effectiveness of combination use of Rimegepant plus NSAIDs/Triptans/Combination analgesic in participants with insufficient response to monotherapy.
* To evaluate the acute treatment effectiveness of Rimegepant in migraine participants with prior treatment failure of more than two triptans.

Study design This is a single arm, prospective, multi-center, observational registry study with participants receiving Rimegepant for the acute treatment of migraine in a real-world setting. Each participant will receive treatment and care according to standard clinical practice.

About 3,000 adult migraine participants will be enrolled continuously at 70 to 73 sites with a headache clinic or headache center in China in approximately 16 consecutive months or until reaching the target sample size.. The index date for a participant will be the date of enrollment. The maximum follow-up period per participant after enrollment is 12 months.

At the Baseline Visit, the demographics information, socioeconomic characteristics, and medical and migraine history will be collected from the enrolled participants. For the acute treatment effectiveness evaluation, data on Rimegepant treating single migraine attack including the timing of dosing, most severe pain, onset time of pain relief, onset time of associated symptoms relief, satisfaction with pain relief and satisfaction with function improvement are expected to be captured within 3 months after enrollment through a digital platform. If none of these data are captured within 3 months, the participant will be marked as failed in the study and will not be followed up further. For the long-term effectiveness evaluation, participants will use an eDiary to record headache and migraine occurrence, and use a digital platform to collect Rimegepant and other migraine-related medication usage days every month. At study visits, participants will complete the Migraine-Specific Quality-of-Life Questionnaire (MSQ) v2.1, Migraine Disability Assessment (MIDAS), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder -7 (GAD-7), Patient Global Impression of Change (PGI-C) and the Satisfaction with Medication (SM) scale at months 3, 6 and 12 via electronic patient reported outcomes (ePROs). The previous four scales will be completed by participants at baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be eligible for inclusion in the study:

  1. Male or female participants aged ≥ 18 years-old
  2. Primary diagnosis of migraine according to ICHD-3
  3. Migraine attacks present for more than 1 year
  4. Rimegepant is prescribed for the acute treatment of migraine by physician
  5. Written informed consent must be obtained before participant is enrolled

Exclusion Criteria:

* Participants meeting any of the following criteria will not be included in the study:

  1. Severe impairment of speech, vision, memory or cognition, or other factors that affect communication and ability to complete questionnaires and follow-up
  2. Lack of necessary digital tools to complete questionnaires on a digital platform
  3. History of hypersensitivity reaction to Rimegepant or to any of its components
  4. Participants with severe hepatic impairment or end-stage renal disease
  5. Any situation that the investigator believes may affect the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit male and female participants in China, 18 years of age or older with migraine (with or without aura), diagnosed according to the International Classification of Headache Disorders, 3rd edition (ICHD-3)21. Participants must be prescribed with Rimegepant according to the clinical decision of the doctor and the willingness of the participants.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
The average scores of the most severe pain post-dose measured by VAS scale to evaluate the effectiveness of Rimegepant in the acute treatment of migraine | within 48 hours post-dose of rimegepant
  Pain severity post-dose will be measured on Visual Analogue Scale (VAS) (0=No pain, 10=worst pain).
The onset time of pain relief post-dose to evaluate the effectiveness of Rimegepant in the acute treatment of migraine | within 48 hours post-dose of rimegepant
  Onset of pain relief is defined as the earliest time point after dosing at which the participant feels that the medication has started working to relieve the pain. If the participant remains pain free both at and after dosing, the time should be recorded as 0
The percentage of patients satisfied with pain relief post-dose to evaluate the effectiveness of Rimegepant in the acute treatment of migraine | within 48 hours post-dose of rimegepant
  Satisfaction with pain relief will be measured via 7-point SM scale
The percentage of patients satisfied with return to normal function post-dose to evaluate the effectiveness of Rimegepant in the acute treatment of migraine | within 48 hours post-dose of rimegepant
  Satisfaction with pain relief will be measured via 7-point SM scale

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhenjiang

IPD SHARING:
Plan to Share IPD: No